CLINICAL TRIAL: NCT06552299
Title: Evaluating Length and Depth Estimation Accuracy
Brief Title: Evaluating Length and Depth Estimation Accuracy of Laypersons and Health-Care Providers
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Collaborators: SMG-SNU Boramae Medical Center (Other)
Responsible Party: Principal Investigator, Stephen Gyung Won Lee, Assistant professor, SMG-SNU Boramae Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 30-2024-42
Record Dates: First submitted 2024-08-11; First posted 2024-08-14 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2025-01

CONDITIONS: Cardiopulmonary Resuscitation
Keywords: Cardiopulmonary Resuscitation; Cardiac Arrest
MeSH Terms: conditions — Heart Arrest | interventions — Health Personnel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Laypersons (Experimental): Adult laypersons without cardiopulmonary resuscitation training within 2 years.
  Interventions: Other: Laypersons
- Health-Care Providers (Active Comparator): Adult health-care providers (doctors, nurses and emergency medical technicians).
  Interventions: Other: Health-Care Providers

INTERVENTIONS:
Other: Laypersons — 1. Participants will be asked to draw a 5cm line.
  2. Participants will be asked to press a depth measuring device and resuscitation training manikin to depth of 5cm without and with assistance.
  Arms: Laypersons
Other: Health-Care Providers — 1. Participants will be asked to draw a 5cm line.
  2. Participants will be asked to press a depth measuring device and resuscitation training manikin to depth of 5cm without and with assistance.
  Arms: Health-Care Providers

SUMMARY:
The objective of the study is to measure accurateness of length and depth estimation of laypersons and health-care providers.

DETAILED DESCRIPTION:
The study hypothesis is that both laypersons and health-care providers will have difficulty estimating length and depth. The study will enroll 100 laypersons and 100 health-care providers. The participants will be asked to draw a 5cm line without assistance an estimate 5cm depth to measure accurateness of length and depth estimation.

ELIGIBILITY:
Inclusion criteria:

* Laypersons: adult laypersons without cardiopulmonary resuscitation training within 2 years
* Health-care providers: adult health-care providers (doctors, nurses and emergency medical technicians)

Exclusion criteria:

* Laypersons: laypersons with cardiopulmonary resuscitation training within 2 years.
* Health-care providers: health-care providers who are inactive (not currently working at medical facilities)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-08-27 (Actual); Primary Completion 2025-01-05 (Actual); Study Completion 2025-02-25 (Estimated)

PRIMARY OUTCOMES:
Depth estimation | Measurement immediately after registration on the day of arrival at the study site (protocol will take less than 5 minutes to complete)
  Depth pressed by participants measured by depth measuring device

SECONDARY OUTCOMES:
Length estimation | Measurement immediately after registration on the day of arrival at the study site (protocol will take less than 5 minutes to complete)
  Length of line drawn by participants
Depth estimation with assistance | Measurement immediately after registration on the day of arrival at the study site (protocol will take less than 5 minutes to complete)
  Depth pressed by participants measured by depth measuring device with assistance

CONTACTS AND LOCATIONS:
Overall Officials: STEPHEN GW LEE, MD, MA, Principal Investigator — SMG-SNU Boramae Medical Center
Locations (1):
- SMG-SNU Boramae Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Panchal AR, Bartos JA, Cabanas JG, Donnino MW, Drennan IR, Hirsch KG, Kudenchuk PJ, Kurz MC, Lavonas EJ, Morley PT, O'Neil BJ, Peberdy MA, Rittenberger JC, Rodriguez AJ, Sawyer KN, Berg KM; Adult Basic and Advanced Life Support Writing Group. Part 3: Adult Basic and Advanced Life Support: 2020 American Heart Association Guidelines for Cardiopulmonary Resuscitation and Emergency Cardiovascular Care. Circulation. 2020 Oct 20;142(16_suppl_2):S366-S468. doi: 10.1161/CIR.0000000000000916. Epub 2020 Oct 21. No abstract available. PMID 33081529
- [Background] Olasveengen TM, Semeraro F, Ristagno G, Castren M, Handley A, Kuzovlev A, Monsieurs KG, Raffay V, Smyth M, Soar J, Svavarsdottir H, Perkins GD. European Resuscitation Council Guidelines 2021: Basic Life Support. Resuscitation. 2021 Apr;161:98-114. doi: 10.1016/j.resuscitation.2021.02.009. Epub 2021 Mar 24. PMID 33773835
- [Background] van Tulder R, Laggner R, Kienbacher C, Schmid B, Zajicek A, Haidvogel J, Sebald D, Laggner AN, Herkner H, Sterz F, Eisenburger P. The capability of professional- and lay-rescuers to estimate the chest compression-depth target: a short, randomized experiment. Resuscitation. 2015 Apr;89:137-41. doi: 10.1016/j.resuscitation.2015.01.031. Epub 2015 Feb 4. PMID 25660952
- [Background] Trethewey SP, Vyas H, Evans S, Hall M, Melody T, Perkins GD, Couper K. The impact of resuscitation guideline terminology on quality of dispatcher-assisted cardiopulmonary resuscitation: A randomised controlled manikin study. Resuscitation. 2019 Sep;142:91-96. doi: 10.1016/j.resuscitation.2019.07.016. Epub 2019 Jul 19. PMID 31330198
- [Background] Deakin CD, Sidebottom DB, Potter R. Can rescuers accurately deliver subtle changes to chest compression depth if recommended by future guidelines? Resuscitation. 2018 Mar;124:58-62. doi: 10.1016/j.resuscitation.2018.01.010. Epub 2018 Jan 5. PMID 29309883
- [Background] Mirza M, Brown TB, Saini D, Pepper TL, Nandigam HK, Kaza N, Cofield SS. Instructions to "push as hard as you can" improve average chest compression depth in dispatcher-assisted cardiopulmonary resuscitation. Resuscitation. 2008 Oct;79(1):97-102. doi: 10.1016/j.resuscitation.2008.05.012. Epub 2008 Jul 17. PMID 18635306